CLINICAL TRIAL: NCT03066466
Title: Randomized Study of Atorvastatin Prophylaxis as a Supplement to Standard of Care Prophylaxis to Prevent Chronic Graft Versus Host Disease Allogeneic Stem Cell Transplantation From Matched Unrelated Donors
Brief Title: Randomized Study: Standard of Care With or Without Atorvastatin for Prevention of GVHD for Matched Unrelated Donor BMT
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No participants were enrolled
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Patrick Stiff, Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 208106
Record Dates: First submitted 2017-02-23; First posted 2017-02-28 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Myelodysplastic Syndrome
Keywords: Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Myelodysplastic Syndrome; BMT; Matched unrelated donor transplant; Graft versus Host Disease; GVHD
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Graft vs Host Disease | interventions — Atorvastatin; Methotrexate; Tacrolimus

STUDY DESIGN:
Intervention Model Description: Randomized, two arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Atorvastatin (Experimental): The preventative atorvastatin treatment 40mg daily by mouth for GVHD will start at 14 days prior to transplant & continue until 365 days post-transplant or if significant adverse events occur. Patients will also receive our standard of care for graft versus host disease prevention which consists of two drugs, Methotrexate and Tacrolimus. For all matched unrelated donor allogeneic transplantation patients, the following schedule of Methotrexate 5mg/metered square will be administered IV post-transplant on Days 1, 3 & 6. Tacrolimus will be administered 2 days prior to transplant & continue approximately 180 days post-transplant. Tacrolimus 0.03 mg/kg daily will be administered IV until patient can take it by mouth.
  Interventions: Drug: Atorvastatin; Drug: Methotrexate; Drug: Tacrolimus
- Arm B: Standard of Care (Active Comparator): Patients will receive our standard of care for graft versus host disease prevention which consists of two drugs, Methotrexate and Tacrolimus. For all matched unrelated donor allogeneic transplantation patients, the following schedule of Methotrexate 5mg/metered square will be administered IV post-transplant on Days 1, 3 & 6. Tacrolimus will be administered 2 days prior to transplant & continue approximately 180 days post-transplant. Tacrolimus 0.03 mg/kg daily will be administered IV until patient can take it by mouth.
  Interventions: Drug: Methotrexate; Drug: Tacrolimus

INTERVENTIONS:
Drug: Atorvastatin — Oral medication given to prevent graft versus host disease in bone marrow transplant.
  Other Names: Lipitor
  Arms: Arm A: Atorvastatin
Drug: Methotrexate — IV medication given to prevent graft versus host disease in bone marrow transplant.
  Other Names: Trexall
Drug: Tacrolimus — IV or Oral medication given to prevent graft versus host disease in bone marrow transplant.
  Other Names: Prograft

SUMMARY:
Chronic Graft Versus Host Disease (GVHD) is one of the most challenging complications in long term survivors of allogeneic stem cell transplantation. As the number of allogeneic stem cell transplantations rises annually, the incidence of chronic GVHD rates have also increased due to a variety of factors including but not limited to increasing use of peripheral blood stem cell (PBSC) grafts, increasing age of both donors and recipients, and increased use of matched unrelated donors. One study showed much lower than traditional acute GHVD rate and chronic GHVD which is similar with historical rates when atorvastatin was administered prophylactically to both the donors as well as recipients of matched related allogeneic stem cell transplantation, lead to the interest in further examining the role of Atorvastatin in relation to the development of GVHD. The investigator hypothesize that the administration of atorvastatin in recipients of matched unrelated allogeneic stem cell transplantation, a group with known higher incidence of chronic GHVD, would be a safe and effective method to reduce the incidence of chronic GVHD. Matched related allogeneic stem cell transplantation recipients will not be included in this study due to their significantly lower GVHD rates. The definition and monitoring of our primary endpoint of GVHD is well established in clinical trials in allogeneic stem cell transplantations and the investiagor will utilize the National Institutes of Health (NIH) Staging System for the diagnosis and severity assessment of chronic GVHD as well the recommendations from the NIH Consensus Conference for the conduct of clinical trials in chronic GVHD.

Several secondary endpoints will be examined as defined below and include standard complementary data in the examination of clinical trials in chronic GVHD again as laid out by the NIH Consensus Conference for conduct of clinical trials in chronic GHVD.

DETAILED DESCRIPTION:
This is a randomized, open label phase III trial in patients with Acute Myeloid Leukemia, Acute Lymphocytic Leukemia, and Myelodysplastic Syndrome undergoing matched unrelated donor transplant.

Patients randomized to the treatment arm (atorvastatin):

The prophylaxis atorvastatin treatment (taken by mouth) for GVHD will start at 14 days prior to transplant and continue until 365 days post-transplant or until development of significant adverse events or desire of the primary treating physician to stop the administration.

The patients will also receive our institution's standard graft versus host disease prophylactic regimen which consists of two drugs. It has been shown that immunosuppression with two drugs is better than a single agent thus our institution utilizes a combination of Methotrexate and Tacrolimus. For all matched unrelated donor allogeneic transplantation patients, the following schedule of Methotrexate will be administered intravenously (IV) post-transplant on Days 1, 3 and 6. Tacrolimus will be administered 2 days prior to transplant and continue approximately 180 days post-transplant. Tacrolimus will be administered IV until patient can take it by mouth.

Patients randomized to standard of care:

Patients will receive our institution's standard graft versus host disease prophylactic regimen which consists of two drugs. It has been shown that immunosuppression with two drugs is better than a single agent thus our institution utilizes a combination of Methotrexate and Tacrolimus. For all matched unrelated donor allogeneic transplantation patients, the following schedule of Methotrexate will be administered intravenously (IV) post-transplant on Days 1, 3 and 6. Tacrolimus will be administered 2 days prior to transplant and continue approximately 180 days post-transplant. Tacrolimus will be administered IV until patient can take it by mouth.

ELIGIBILITY:
Inclusion Criteria

* Men or women between 18-65 years of age
* Patients designated to undergo allogeneic peripheral blood or bone marrow stem cell transplantation from matched unrelated donor following the diagnosis of one of the following primary diseases in early or intermediate disease status:

  * AML at the following stages at time of screening: 1st remission, 2nd remission, and 3rd or subsequent remission
  * ALL at the following stages at time of screening: 1st remission, 2nd remission, and 3rd or subsequent remission
  * MDS
* Patients must have Performance Score (PS) greater than 70 percent

Exclusion Criteria

* Cardiac: ejection fraction less than 40 percent or other significant cardiac disease
* Pulmonary: FEV1 or DLCO less than 45 percent
* Renal: creatinine greater than the upper limit of normal
* Hepatic: bilirubin greater than 2.0 times the upper limit of normal
* CNS: documented active CNS disease
* Patients who are known to be positive for Hepatitis B surface antigen or Hepatitis C antibody, or who have tested positive for HIV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-10 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to determine the cumulative incidence of chronic GVHD at one year after stem cell transplantation and treatment with atorvastatin | 2 years
  National Institutes of Health Chronic Graft-Versus-Host Disease Grading and Form

SECONDARY OUTCOMES:
To determine the cumulative incidence of grade 3 to 4 acute GVHD | 100 days
  National Institutes of Health Acute Graft-Versus-Host Disease Grading and Form
To determine rate of disease relapse | 2 years
  Blood work and/or bone marrow biopsy will be used
To determine non-relapse mortality (NRM) | 2 years
  Blood work and/or bone marrow biopsy will be used
To determine progression-free survival (PFS) | 2 years
  Blood work and/or bone marrow biopsy will be used
To determine overall survival (OS) | 2 years
  Blood work and/or bone marrow biopsy will be used
Number of participants with Grade 4 through 5 Adverse Events that are related to study treatment, grading according to NCI CTCAE Version 4 | 30 days of the last dose of protocol treatment
  Toxicities that are possibly, probably, and definitely related
Determine the frequency and severity of chronic GVHD | 2 years
  National Institutes of Health Chronic Graft-Versus-Host Disease Grading and Form

OTHER OUTCOMES:
To determine the effect of atorvastatin on immune reconstitution | 2 years
  Blood work will be used to evaluate recovery of white blood cells, red blood cells and platelets plus T and B cell count subset.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stiff, MD, Study Director — Cardinal Bernardin Cancer Center, Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No